CLINICAL TRIAL: NCT04756128
Title: Impact of Colchicine and Low-dose Naltrexone on COVID-19 Disease Progression and Clinical Course in Hospitalized Patients
Brief Title: Impact of Colchicine and Low-dose Naltrexone on COVID-19
Acronym: COLTREXONE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Park Nicollet Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: X2103400
Record Dates: First submitted 2021-01-28; First posted 2021-02-16 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; Naltrexone; vivitrol

STUDY DESIGN:
Intervention Model Description: This will be a four arm, prospective, randomized, open label trial in patients hospitalized with moderate COVID-19. Randomization will be stratified by baseline severity score (2 or 3) to ensure balanced baseline severities between the four arms. Block randomization will be used to ensure equal group sizes. As the final sample size is unknown, study staff will use small blocks of eight for randomization. This is being done in an effort to ensure evenly distributed treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Colchicine-Only Arm (Experimental): Patients randomized to a colchicine-containing treatment arm will receive colchicine 0.6 mg twice daily for up to 28 days. On the day of enrollment, provided the first dose can be given prior to 16:00 that day, patients are eligible to receive two doses; the second dose will be scheduled for 22:00. Patients experiencing gastrointestinal side effects (nausea, vomiting, and diarrhea) on twice daily dosing may have the dose decreased to 0.6 mg daily. Dosing will continue twice daily unless there is a change that requires a dose adjustment or an exclusion criterion is met. Dosing deviations above the study protocol will be allowed if medically necessary for the treatment of an additional indication (e.g. colchicine for viral pericarditis).
  Patients in this arm will also receive the investigating institution's current standard of care (described in detail in the "standard of care" arm) for patients with COVID-19.
  Interventions: Drug: Colchicine 0.6 mg
- Colchicine and Naltrexone ("Combined") Arm (Experimental): Patients randomized to a colchicine-containing treatment arm (including the "combined arm") will receive colchicine 0.6 mg twice daily for up to 28 days. On the day of enrollment, provided the first dose can be given prior to 16:00 that day, patients are eligible to receive two doses; the second dose will be scheduled for 22:00.
  Patients in the "combined" arm will also receive naltrexone. Patients randomized to an LDN-containing treatment arm (including the "combined arm") will receive naltrexone 4.5 mg once daily. The first dose can be given at any time during the day of enrollment/randomization, and will be timed at 08:00 daily thereafter (with AM colchicine dose, if in combined colchicine/LDN arm) for up to 28 days (unless new contraindication or exclusion criteria met).
  Patients in this arm will also receive the investigating institution's current standard of care (described in detail in the "standard of care" arm) for patients with COVID-19.
  Interventions: Drug: Colchicine 0.6 mg; Drug: Naltrexone
- Naltrexone-Only Arm (Experimental): Patients randomized to an LDN-containing treatment arm (including the "combined arm") will receive naltrexone 4.5 mg once daily. The first dose can be given at any time during the day of enrollment/randomization, and will be timed at 08:00 daily thereafter (with AM colchicine dose, if in combined colchicine/LDN arm) for up to 28 days (unless new contraindication or exclusion criteria met).
  Patients in this arm will also receive the investigating institution's current standard of care (described in detail in the "standard of care" arm) for patients with COVID-19.
  Interventions: Drug: Naltrexone
- Standard of Care Arm (No Intervention): Patients in this arm will receive the investigating institution's current standard of care for patients with COVID-19. For example, all patients requiring supplemental oxygen (assuming no contraindications) would be candidates for both remdesivir 200 mg x 1 IV dose followed the next day by 100 mg q24h IV x up to 4 doses, as well as dexamethasone 6 mg q24h x 10 up to 10 doses.

INTERVENTIONS:
Drug: Colchicine 0.6 mg — Colchicine is an oral anti-inflammatory agent that is relatively inexpensive, readily available, and has been used for generations. Approved for treatment and prophylaxis of gout flares and Mediterranean fever, it is also used in a variety of other inflammatory conditions (e.g. pericarditis and diffuse vascular inflammation such as Behcet syndrome). Colchicine binds to tubulin causing depolymerization, which interferes with neutrophil chemotaxis, adhesion, and mobilization to sites of inflammation, and contributes to reduction in superoxide production; through interference of the NLRP3 inflammasome protein complex, colchicine inhibits IL-1b, IL-6, and IL-18 production.
  For this study, patients enrolled in a colchicine containing arm will receive 0.6mg of colchicine BID (unless renal function/gastrointestinal issues require adjustments described in the protocol)
  Other Names: Colcrys
  Arms: Colchicine and Naltrexone ("Combined") Arm; Colchicine-Only Arm
Drug: Naltrexone — Most well known as an opioid antagonist, or a treatment for alcohol dependence, naltrexone also possesses immunomodulatory effects. Seen exclusively at low doses, this attribute is being employed in the pain community as a novel anti-inflammatory agent that has been shown to reduce symptom severity in fibromyalgia, Crohn's disease, multiple sclerosis, and complex regional pain syndrome.
  For this study, patients enrolled in a naltrexone-containing arm will take their daily dose of the medication (4.5mg) by oral suspension.
  Other Names: Vivitrol
  Arms: Colchicine and Naltrexone ("Combined") Arm; Naltrexone-Only Arm

SUMMARY:
The purpose of this study is to explore the impact of two medications-colchicine and low-dose naltrexone (LDN)-relative to standard of care (SOC) on COVID-19 disease progression to severe/critical illness and/or intubation in patients hospitalized with moderate COVID-19. As researchers have learned, COVID-19's clinical course suggests that the hyperinflammatory response seen in severe/critical cases is involved in the pathogenesis of associated adverse sequelae such as acute respiratory distress syndrome (ARDS), thromboembolic disease, and acute cardiac injury. Given colchicine has demonstrated clinical utility in inflammatory syndromes within these systems (e.g. endothelial/vascular/myocardial), and LDN acts both to boost the immune system, and limit an excessive response; they may prove useful in minimizing the risk of disease progression and associated adverse sequelae.

DETAILED DESCRIPTION:
In December 2019, a novel coronavirus caused a cluster of pneumonia cases in Wuhan, China. The identified virus was officially named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and the associated illness named coronavirus disease (COVID-19) (WHO). In the months since its discovery, the spread of SARS-CoV-2 has led to tens of millions of cases worldwide. In the United States alone, there have been over 11.6 million cases of COVID-19, with over 340,000 attributed deaths reported as of December 31, 2020 (CDC Cases in the US). Despite the recent availability of a preventative vaccine, there are limited pharmacotherapeutic treatment options for those with an active infection, the majority of which remain investigational.

Common symptoms among patients with mild disease include fever, altered senses of smell or taste, fatigue, or cough. More severe cases of COVID-19 may lead to hypoxemia and pneumonia. When compared to those with less-severe disease, severe/critical COVID-19 pneumonia generally results in an increase in circulating proinflammatory chemokines and cytokines. The SARS-CoV-2 virus has specific structural components (e.g. viroporin E and viroporins 3a and 8A) that have been shown to activate NLRP3 inflammasomes NLRP3 has been found to be a major pathophysiologic component in developing ARDS; and inflammasome activation along with subsequent cytokine production is seen with myocardial injury, which may provide mechanistic insight to SARS-CoV-2's ability to cause cardiac insult. Additionally, aberrant activation of neutrophils and formation of excessive neutrophil extracellular traps (NETs) were found to be associated with ARDS, and recently to be the potential central cause of severe/critical COVID-19.

Treatments that influence neutrophil recruitment to sites of inflammation and hyper-inflammatory response may prove beneficial for reduction in disease progression, adverse sequelae, and mortality associated with COVID-19 infections. Agents under investigation to mitigate this detrimental host response include the IL-6 receptor antagonists. However, their extreme expense, scarce availability, and high-risk for severe adverse effects relegate the use of these injectable agents to cases that have already progressed to critical illness.

Colchicine is an oral anti-inflammatory agent that is relatively inexpensive, readily available, and has been used for generations. Approved for treatment and prophylaxis of gout flares and Mediterranean fever, it is also used in a variety of other inflammatory conditions. Colchicine binds to tubulin causing depolymerization, which interferes with neutrophil chemotaxis, adhesion, and mobilization to sites of inflammation, and contributes to reduction in superoxide production; through interference of the NLRP3 inflammasome protein complex, colchicine inhibits IL-1b, IL-6, and IL-18 production. These are recognized as playing an important role in acute coronary syndrome, pericarditis, and ARDS. Colchicine also has an anti-apoptotic action on endothelial cells that may provide benefit in minimizing extravasation, capillary leak, and therefore progression or development of ARDS. Lastly, coronavirus replication, virion particle assembly, and subsequent exocytosis from the host cell, have been shown to rely on cytoplasmic structural proteins (microtubules) for trafficking during its lifecycle. Disrupting microtubule trafficking has the potential to interfere with these key viral replication steps, and therefore introduction of a microtubule depolymerizing agent may help treat a coronavirus infection through decreased viral replication.

The use of colchicine in patients hospitalized with COVID-19 has been studied in several small uncontrolled case series and comparative cohort studies, as well as small, randomized controlled trials. Results have been unanimously favorable thus far, though they have substantial limitations. Some were performed during local COVID-19 surges, rates of intubation and mortality were likely inflated as a result, and therefore the benefits of colchicine may be overestimated.

Most well known as an opioid antagonist, or a treatment for alcohol dependence, naltrexone also possesses immunomodulatory effects. Seen exclusively at low doses, this attribute is being employed in the pain community as a novel anti-inflammatory agent that has been shown to reduce symptom severity in fibromyalgia, Crohn's disease, and multiple sclerosis. Naltrexone is a 50:50 racemic mixture of both L and R isomers - in theory, these isomers allow it to act in a dualistic fashion, both boosting the immune system yet limiting an excessive immune response. The L isomer is a competitive inhibitor of the Mu and Kappa opioid receptor, resulting in elevated levels of endogenous endorphins and enkephalins, which in turn, functions as an immune enhancer. The R isomer blocks the toll like receptor and modulates T and B cell activity; the downstream effects limit the release of inflammatory cytokines including IL-6, IL-12, TNF alpha, and NF-KB. A study in 2017 demonstrated a significant reduction in cytokines after eight weeks of therapy in eight female patients.

While preliminary LDN studies demonstrate success in Crohn's disease, multiple sclerosis, and fibromyalgia, there is still a need for follow-up trials to establish definitive evidence of benefit. The lack of proprietary value in a generic medication with no industry backing has hampered widespread adoption and FDA approval. Thus, clinical efficacy data is slowly forthcoming on LDN. At the same time, the safety profile of naltrexone is well established and very well tolerated in alcohol use disorder. Considering that is a high-risk population, and the dose used is significantly higher (25-100mg versus 1-4.5mg for LDN), it stands to reason that LDN should have little to no toxicity. Hepatic function has to be monitored at higher doses, and the drug should be stopped if necessary. However, with LDN the majority of adverse drug effects are constitutional (headache, dizziness, nausea etc.), with no end organ damage and no evidence for opportunistic infections.

As previously outlined, available evidence demonstrates that excessive immune response in the form of a "cytokine storm" plays a key role in the pathophysiology of COVID-19 offering this process as a possible target for drug therapy. Known immunomodulatory effects of LDN suggest that this drug could be used to reduce this exaggerated immune response. While the efficacy of LDN is being studied in COVID-19 (NCT04604704, NCT04604678, NCT04365985) in combination with a nutritional supplement, metformin, and ketamine (respectively), only the latter trial is recruiting at this time, and none includes colchicine.

The proposed study will investigate whether or not the colchicine and naltrexone (used alone or in combination) can slow the progression of COVID-19 patients hospitalized with mild illness. A modified version of the World Health Organization's R&D Blueprint Ordinal Clinical Scale will be used to assess this outcome. Patients enrolled in the study will follow the schedule of events outlined below. If randomized to receive study drug (colchicine only, naltrexone only, or both colchicine and naltrexone) patients will continue to take the medication until discharge form the hospital (but not more than 28 days).

Baseline Enrollment Information collection

* Inclusion & Exclusion Criteria Assessment
* Informed consent, randomization
* Demographics-Documentation of patient characteristics
* Past medical history-Documentation of diagnoses at baseline
* Documentation of need for supplemental home oxygen therapy at baseline
* Rule out pregnancy for female participants of child-bearing age Clinical Course Monitoring - Performed daily until discharge
* Safety assessment and reporting-Review of chart for AEs by study staff
* Concomitant medications-Review of medications taken in hospital in addition to study drugs
* New Drug-Drug Interactions-Assessment of new/updated medications to determine risk of new drug interactions
* Documentation of Colchicine dose frequency (Daily/BID, with rationale if changed)
* Study Drug Administration-For interventional arms: Documentation of date and time of study drug administration
* Maximum O2 needs for continuous 12-hour periods beginning at hospital admission
* Tmax-Maximum recorded temperature patient reached during the study day
* Chest imaging (yes/no)-Documentation of whether patient received SOC chest imaging on study day
* EKG or continuous telemetry (yes/no)-Documentation of whether patient received an SOC EKG or is on continuous telemetry on study day
* LMWH > 0.5 mg/kg/dose (not cumulative daily dose) or heparin drip? (yes/no)-Documentation of need for more than .5mg/kg total dose of Low Molecular Weight Heparin on study day
* Level of care-Documentation of clinical scale score; hospital unit through which patient is being treated
* Length of hospitalization Mortality-Documentation of patient death at any time during the hospital stay Laboratory Monitoring
* BNP (B-Type Natriuretic Peptide)-Documented during patient's hospital stay as performed per SOC
* CBC with differential-Documented during patient's hospital stay as performed per SOC with supplemental research-only labs added as needed
* C-reactive protein-Documented during patient's hospital stay as performed per SOC with supplemental research-only labs added as need
* D-dimer-Documented during patient's hospital stay as performed per SOC with supplemental research-only labs added as need
* Ferritin-Documented during patient's hospital stay as performed per SOC with supplemental research-only labs added as need
* Hepatic Function Panel-Documented during patient's hospital stay as performed per SOC with supplemental research-only labs added as need
* Procalcitonin-Documented during patient's hospital stay as performed per SOC -Serum Creatinine (SCr)-Documented during patient's hospital stay as preformed per SOC/as needed for research
* Troponin-Documented during patient's hospital stay as performed per SOC up to discharge

Dosing strategy-Colchicine Patients randomized to a colchicine-containing treatment arm will receive colchicine 0.6 mg twice daily for up to 28 days. On the day of enrollment, provided the first dose can be given prior to 16:00 that day, patients are eligible to receive two doses; the second dose will be scheduled for 22:00. Patients experiencing gastrointestinal side effects (nausea, vomiting, and diarrhea) on twice daily dosing may have the dose decreased to 0.6 mg daily. Dosing will continue twice daily unless there is a change that requires a dose adjustment or an exclusion criterion is met. Dosing deviations above the study protocol will be allowed if medically necessary for the treatment of an additional indication (e.g. colchicine for viral pericarditis).

Renal dosing:

* CrCl* ≥50 mL/min: colchicine 0.6 mg twice daily
* CrCl* 30-49 mL/min: colchicine 0.6 mg every 24 hours
* CrCl* 11-29 mL/min**: colchicine 0.6 mg every 48 hours
* CrCl* ≤10 mL/min: doses will be held

Drug interactions: To ensure patients are properly screened and identified as eligible/ineligible with respect to prescribed medications, this research team will identify a group of study pharmacists and physicians (including the PI, Dr. Daniel Delaney, and a pain specialist, Dr. Joseph Johnson), who will be available as-needed to field questions regarding any medications a patient is taking during or prior to their hospital stay that may or may not preclude study participation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and (non-pregnant, non-breastfeeding) females aged 18 years or older
2. Requiring admission to Methodist or Regions Hospital due to laboratory-confirmed COVID-19
3. Meets criteria of only up to moderate COVID-19 disease as defined by a clinical score of 2 or 3 at the time of enrollment, and one or more of the following:

   1. Dyspnea limiting usual activities on baseline O2 needs
   2. Respiratory rate >/= 30/min on O2 or room air
   3. Blood oxygen saturations <94% on room air (or on baseline O2 needs if on supplemental oxygen prior to presentation at the hospital for a condition unrelated to COVID-19).
   4. Requiring supplemental 02 above baseline needs (i.e. prior to presentation at hospital)
   5. COVID-19 contributed to the current hospital admission, per attending provider's clinical assessment of the patient.
4. Ability to provide written informed consent, or has identifiable LAR that is able to do so on the patient's behalf as defined by study protocol, prior to performing study procedures.

Exclusion Criteria:

1. Patients meeting criteria for severe/critical COVID-19 as defined by study protocol or requiring O2 supplementation ≥10L nasal cannula at screening
2. Patients currently in shock as defined by hemodynamic instability requiring vasopressors
3. Patients with a current hospitalization for COVID-19 that is >/=7 days at the time of screening.
4. Clinical estimation of attending physician that the patient will require mechanical respiratory support within 48 hours of enrollment
5. Patients in which EITHER symptom onset OR a positive COVID-19 laboratory test occurred >14 days prior to enrollment.
6. Patients with concomitant influenza A or B at time of hospitalization if tested as part of ED/hospital admission.
7. Female patients who are pregnant or breastfeeding at time of hospital admission
8. Diagnosis of Chronic Kidney Disease stage ≥4 as documented in the patient's problem list (not based on CrCI calculations alone)
9. CrCl < 30 mL/min or requiring renal replacement therapy (e.g. intermittent hemodialysis, continuous renal replacement therapy, peritoneal dialysis) at screening
10. History of cirrhosis or advanced liver disease, or active hepatic viral infection
11. Transplant of kidney, lung, heart, or liver in the past 2 years
12. Uncontrolled severe gastrointestinal disorders, Crohn's disease, ulcerative colitis, chronic diarrhea, diarrhea predominant irritable bowel syndrome, active stomach or intestinal ulcer, or one that was treated within the last 6 months
13. Patients currently receiving agents that are p-glycoprotein AND strong CYP3A4 inhibitors with CrCl < 60 mL/min, or any combination of drug interactions that is not amenable to dosage adjustment (refer to list of medications with potential Colchicine and Naltrexone interactions).
14. Patients actively undergoing chemotherapy for an active malignancy, or history of a hematologic malignancies
15. Chronic or current use of colchicine or any mu-opioid antagonist.
16. Chronic, scheduled opioid therapy (i.e. not intermittent as needed use), or, prior to enrollment, an acute condition requiring continued pain control that is unattainable without ongoing opioid therapy.
17. Pre-existing condition that is being treated with tocilizumab, anakinra, sarilumab, other interleukin-antagonists, TNF-inhibitors, or JAK inhibitors.
18. NOTE: Patients treated with tocilizumab will be permitted to enroll if their care team is prescribing it for COVID-19. Use of tocilizumab at baseline for another indication will continue to be excluded.
19. Participation in any other clinical trial of an experimental treatment for COVID-19, note:

    1. While convalescent plasma is no longer recommended within HP, it can be given if deemed appropriate by the medical team once ≥ 24 hours has elapsed since enrollment;
    2. Patients previously enrolled in the C3PO study can enroll in this study, as any convalescent plasma received would have been outpatient;
    3. Remdesivir is allowed per standard protocol;
    4. Dexamethasone is allowed per standard protocol
20. Patients actively enrolled in hospice or that are DNI or on palliative care
21. History of hypersensitivity reaction to colchicine or its inactive ingredients
22. History of hypersensitivity reaction to naltrexone or its inactive ingredients
23. Incarcerated or a ward of the state
24. Any patient considered an unsuitable candidate, for any reason, by study investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-11-26 (Actual); Study Completion 2021-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Delaney, PharmD, Principal Investigator — Park Nicollet Methodist Hospital
Locations (2):
- United States (2):
  - Park Nicollet Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with investigators not currently involved in the study.

RESULTS

PARTICIPANT FLOW:
Groups:
- Colchicine-Only Arm: Patients randomized to a colchicine-containing treatment arm will receive colchicine 0.6 mg twice daily for up to 28 days. Patients experiencing gastrointestinal side effects (nausea, vomiting, and diarrhea) on twice daily dosing may have the dose decreased to 0.6 mg daily. Dosing will continue twice daily unless there is a change that requires a dose adjustment or an exclusion criterion is met. Dosing deviations above the study protocol will be allowed if medically necessary for the treatment of an additional indication (e.g. colchicine for viral pericarditis).
  Patients in this arm will also receive the investigating institution's current standard of care (described in detail in the "standard of care" arm) for patients with COVID-19.
  Colchicine 0.6 mg: Colchicine is an oral anti-inflammatory agent that is relatively inexpensive, readily available, and has been used for generations. Approved for treatment and prophylaxis of gout flares and Mediterranean fever, it is also used in a variety of other inflammatory conditions (e.g. pericarditis and diffuse vascular inflammation such as Behcet syndrome). Colchicine binds to tubulin causing depolymerization, which interferes with neutrophil chemotaxis, adhesion, and mobilization to sites of inflammation, and contributes to reduction in superoxide production; through interference of the NLRP3 inflammasome protein complex, colchicine inhibits IL-1b, IL-6, and IL-18 production.
- Colchicine and Naltrexone ("Combined") Arm: Patients randomized to a colchicine-containing treatment arm (including the "combined arm") will receive colchicine 0.6 mg twice daily for up to 28 days.
  Patients in the "combined" arm will also receive naltrexone. Patients randomized to an LDN-containing treatment arm (including the "combined arm") will receive naltrexone 4.5 mg once daily.
  Patients in this arm will also receive the investigating institution's current standard of care (described in detail in the "standard of care" arm) for patients with COVID-19.
  Colchicine 0.6 mg: Colchicine is an oral anti-inflammatory agent that is relatively inexpensive, readily available, and has been used for generations. Approved for treatment and prophylaxis of gout flares and Mediterranean fever, it is also used in a variety of other inflammatory conditions (e.g. pericarditis and diffuse vascular inflammation such as Behcet syndrome). Colchicine binds to tubulin causing depolymerization, which interferes with neutrophil chemotaxis, adhesion, and mobilization to sites of inflammation, and contributes to reduction in superoxide production; through interference of the NLRP3 inflammasome protein complex, colchicine inhibits IL-1b, IL-6, and IL-18 production.
  Naltrexone: Most well known as an opioid antagonist, or a treatment for alcohol dependence, naltrexone also possesses immunomodulatory effects. Seen exclusively at low doses, this attribute is being employed in the pain community as a novel anti-inflammatory agent.
- Naltrexone-Only Arm: Patients randomized to an LDN-containing treatment arm (including the "combined arm") will receive naltrexone 4.5 mg once daily. The first dose can be given at any time during the day of enrollment/randomization, and will be timed at 08:00 daily thereafter (with AM colchicine dose, if in combined colchicine/LDN arm) for up to 28 days (unless new contraindication or exclusion criteria met).
  Patients in this arm will also receive the investigating institution's current standard of care (described in detail in the "standard of care" arm) for patients with COVID-19.
  Naltrexone: Most well known as an opioid antagonist, or a treatment for alcohol dependence, naltrexone also possesses immunomodulatory effects. Seen exclusively at low doses, this attribute is being employed in the pain community as a novel anti-inflammatory agent that has been shown to reduce symptom severity in fibromyalgia, Crohn's disease, multiple sclerosis, and complex regional pain syndrome.
  For this study, patients enrolled in a naltrexone-containing arm will take their daily dose of the medication (4.5mg) by oral suspension.
Period: Overall Study
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm
Started | 35 | 35 | 36 | 36
Completed | 34 | 33 | 35 | 35
Not Completed | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Total
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11) | 55 (15) | 59 (16) | 59 (16) | 58 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 19 | 16 | 58
  Male | 20 | 24 | 16 | 19 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 0 | 10
  Not Hispanic or Latino | 29 | 30 | 32 | 35 | 126
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 24 | 24 | 24 | 25 | 97
  Black or African American | 3 | 5 | 4 | 7 | 19
  Hispanic | 3 | 2 | 3 | 0 | 8
  Asian | 1 | 1 | 2 | 3 | 7
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Unknown | 2 | 1 | 0 | 0 | 3
  Other | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 34 | 33 | 35 | 35 | 137

OUTCOME MEASURES:

1. Primary Outcome: In Patients Hospitalized With Moderate COVID-19, the Impact of Colchicine and LDN, Alone or in Combination, on Achieving Disease Recovery by Day 5.
Description: Disease recovery from moderate COVID-19 was defined as achieving a clinical scale score of 1 (indicating the patient no longer required hospital-level care for COVID-19. Attainment of a score of 1 by study day 5 was chosen based on initial experience treating COVID-19 within this specific health system-patients with similar disease severity were typically hospitalized for 6-7 days, and time from admission to enrollment in preceding COVID-19 studies was generally 1-2 days.
Time Frame: Assessed from time of hospitalization until (1) 5 days after enrollment, while still hospitalized (or until discharge, which may be less than 5 days)
Measure: Count of Participants; unit: Participants
Groups:
- Colchicine Group: All subjects who received Colchicine from being randomized into Colchicine-Only Arm or Colchicine and Naltrexone Combined Arm
- No Colchicine Group: All subjects who did not receive Colchicine from being randomized into the Naltrexone-Only Arm and Standard of Care Arm
- Naltrexone Group: All subjects who received Naltrexone from being randomized into Colchicine and Naltrexone Combined Arm or Naltrexone-Only Arm
- No Naltrexone Group: All subjects who did not receive Naltrexone from being randomized into the Colchicine-Only Arm and Standard of Care Arm
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 67 | 70 | 68 | 69
Participants | 22 | 24 | 20 | 18 | 46 | 38 | 44 | 40

2. Secondary Outcome: Total Duration of Hospitalization
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on total amount of time (in days) patient spent in hospital from admission to discharge
Time Frame: Assessed from time of hospitalization until discharge, calculated after patient completes hospital stay - approximately 7 days on average
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 67 | 70 | 68 | 69
days | 4.5 [3 to 8] | 4.7 [4 to 6] | 5.7 [3 to 10] | 6.0 [5 to 10] | 4.7 [4 to 7] | 5.7 [4 to 10] | 4.8 [3 to 9] | 4.9 [4 to 10]

3. Secondary Outcome: Total Duration of Hospitalization (From First Dose of Study Drug to Discharge)
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on total amount of time (in days) patient spent in hospital from first dose of any study medication (or when first dose would be given for standard of care arm) to hospital discharge (or when ready for discharge but remains hospitalized for non-medical reasons [e.g. transitional care unit placement delays])
Time Frame: Assessed from time of study drug administration to discharge, calculated after patient completes hospital stay; 7 days after admission on average)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 67 | 70 | 68 | 69
days | 3.5 [2 to 7] | 3.7 [3 to 5] | 4.6 [2 to 8] | 4.3 [3 to 8] | 3.7 [2 to 5] | 4.5 [3 to 8] | 3.8 [2 to 7] | 3.9 [3 to 8]

4. Secondary Outcome: In Patients Hospitalized With Moderate COVID-19, Subjects Who Required Remdesivir
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on requiring remdesivir
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 67 | 70 | 68 | 69
Participants | 20 | 23 | 25 | 24 | 43 | 49 | 48 | 44

5. Secondary Outcome: The Number of Doses of Remdesivir Required In Patients Hospitalized With Moderate COVID-19
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on the number of doses of Remdesivir received. This was only used in patients who met/required this outcome (received Remdesiver, n=92)
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: doses
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 20 | 23 | 25 | 24 | 43 | 49 | 48 | 44
doses | 4.5 [3 to 5] | 4 [2 to 5] | 5 [3 to 5] | 5 [4 to 5] | 4 [3 to 5] | 5 [4 to 5] | 4 [3 to 5] | 5 [3 to 5]

6. Secondary Outcome: In Patients Hospitalized With Moderate COVID-19, Subjects Who Required Corticosteroids
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on requiring corticosteroids
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 67 | 70 | 68 | 69
Participants | 31 | 31 | 34 | 33 | 62 | 67 | 65 | 64

7. Secondary Outcome: The Dosage Amount (in Milligrams) of Corticosteroids Required In Patients Hospitalized With Moderate COVID-19
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on the amount in milligrams (mg) of corticosteroids required. This was only used in patients who met/required this outcome (received Corticosteroids, n=129)
Time Frame: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 31 | 31 | 34 | 33 | 62 | 67 | 65 | 64
mg | 200 [160 to 360] | 200 [147 to 240] | 240 [120 to 360] | 240 [200 to 400] | 200 [160 to 280] | 240 [160 to 400] | 200 [120 to 320] | 233 [160 to 400]

8. Secondary Outcome: In Patients Hospitalized With Moderate COVID-19, The Need for High Flow Nasal Cannula (HFNC) or Non-Invasive Positive Pressure Ventilation (NIPPV)
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on the need of oxygen supplementation with High Flow Nasal Cannula (HFNC) or Non-Invasive Positive Pressure Ventilation (NIPPV)
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 67 | 70 | 68 | 69
Participants | 6 | 8 | 9 | 9 | 14 | 18 | 17 | 15

9. Secondary Outcome: In Patients Hospitalized With Moderate COVID-19, Patients Who Required ICU or ICU Stepdown Cares
Description: Study team will investigate the effects of colchicine and LDN, alone or in combination, on requiring ICU or Stepdown ICU admission
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm | Colchicine Group | No Colchicine Group | Naltrexone Group | No Naltrexone Group
Number analyzed (Participants) | 34 | 33 | 35 | 35 | 67 | 70 | 68 | 69
Participants | 2 | 2 | 6 | 3 | 4 | 9 | 8 | 5

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Colchicine-Only Arm | Colchicine and Naltrexone ("Combined") Arm | Naltrexone-Only Arm | Standard of Care Arm
All-Cause Mortality (participants affected / at risk) | 0/34 | 1/33 | 4/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 4/34 | 6/33 | 6/35 | 3/35
Other Adverse Events (participants affected / at risk) | 13/34 | 19/33 | 13/35 | 14/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colchicine-Only Arm (N=34) | Colchicine and Naltrexone ("Combined") Arm (N=33) | Naltrexone-Only Arm (N=35) | Standard of Care Arm (N=35)
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 — Respiratory failure requiring invasive ventilation
Shock (Cardiac disorders) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Tracheostomy (Surgical and medical procedures) | 1 | 1 | 0 | 0 — Prolonged mechanical ventilation requiring tracheostomy
Parenteral Gastrostomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Transaminitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Deep venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Colchicine-Only Arm (N=34) | Colchicine and Naltrexone ("Combined") Arm (N=33) | Naltrexone-Only Arm (N=35) | Standard of Care Arm (N=35)
Diarrhea/Loose Stools/Incontinence (Gastrointestinal disorders) | 4 | 4 | 2 | 7
Dizziness (General disorders) | 1 | 3 | 0 | 0
Nausea/Stomach Pain/Vomiting (Gastrointestinal disorders) | 4 | 4 | 3 | 1
Anxiety/Agitation (Psychiatric disorders) | 1 | 4 | 4 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 2
Transaminitis (Hepatobiliary disorders) | 2 | 3 | 3 | 3 — Lab results used to determine Transaminitis

LIMITATIONS AND CAVEATS:
Limitations include use of a SOC control in place of placebo given the limited time and resources during the COVID-19 surge. Incidence of disease recovery for both study drugs could be impacted by the rapidly improving standard of care for treating patients as the study progressed (remdesivir, glucocorticoids, and tocilizumab).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT04756128/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT04756128/ICF_000.pdf